CLINICAL TRIAL: NCT01110850
Title: Direct Measurement of Leukemic Cell Turnover (Synthesis and Removal) in Patients With Chronic Lymphocytic Leukemia Using Deuterated Water (GAC 0004)
Brief Title: Direct Measurement of Leukemic Cell Turnover (Synthesis and Removal) in Patients With Chronic Lymphocytic Leukemia (CLL) Using Deuterated Water
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 01-054; GAC # 0004 (Other: GAC # 0004)
Record Dates: First submitted 2009-12-10; First posted 2010-04-27 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Cells, Bone MArrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia: Chronic Lymphocytic Leukemia

SUMMARY:
Chronic lymphocytic leukemia. B-cell chronic lymphocytic leukemia (B-CLL) is the most prevalent leukemia in the Western Hemisphere, accounting for ~25% of all leukemia's. It represents a monoclonal expansion of small, long-lived, apparently slowly dividing CD5+ B cells. Because of the low proliferative index and a presumed uniform proliferative rate of B-CLL cells in vivo (a fact not yet tested or documented), B-CLL appears to be primarily a disease of accumulation rather than proliferation.

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia. B-cell chronic lymphocytic leukemia (B-CLL) is the most prevalent leukemia in the Western Hemisphere, accounting for ~25% of all leukemia's. It represents a monoclonal expansion of small, long-lived, apparently slowly dividing CD5+ B cells. Because of the low proliferative index and a presumed uniform proliferative rate of B-CLL cells in vivo (a fact not yet tested or documented), B-CLL appears to be primarily a disease of accumulation rather than proliferation.

B-CLL remains an incurable illness and there is no survival benefit to early intervention.

Therefore, patients with early stage disease are usually followed closely without initiating treatment. Patients with more extensive disease or progressive cytopenias are eventually treated with cytotoxic agents, with or without prednisone, or with nucleoside analogues that promote apoptosis in the leukemic cells. The clinical outcome of the disease is determined both by the profound dysregulation of the immune system that results in infection and autoimmunity and by leukemic infiltration and destruction of organs. Autoimmune phenomena are common and frequently directed against hematopoietic cells, resulting in autoimmune hemolytic anemia (10-25%) or immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age.
* Must meet the clinical and laboratory criteria for B-CLL (i.e., compatible clinical history and physical exam, presence of lymphocytosis, i.e., >10,000 lymphocytes / mm3, evidence for a monoclonal population of CD5+/CD19+/CD23+ cells in the periphery that have dim surface membrane lg with L chain isotype restriction).
* All patients will be staged according to the system of Rai. Only new onset patients who are not receiving therapy will be entered into the heavy water leukemic cell turnover studies.

Exclusion Criteria:

* Patients hospitalized for an acute medical problem, related or not to their leukemia, within 4 weeks of enrollment.
* A history of a second malignancy involving the hematopoietic system, or the need for extensive chemotherapy for any second malignancy; patients with active immunologic disorders (e.g., HIV and AIDS), especially autoimmune problems (e.g., autoimmune hemolytic anemia of any cause other than B-CLL).
* Patients with impaired decision-making capabilities, e.g. dementia, psychosis, alcoholism, and illicit drug use will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Lymphocytic Leukemia
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2001-06; Primary Completion 2018-05 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
B Cell Chronic Lymphocytic Leukemia Subgroups: Direct measurement of leukemic cell turnover (synthesis and removal) using deuterated water as a DNA-labeling agent in patients with chronic lymphocytic leukemia | 1 year
  We believe that the results of these studies may identify in vivo correlates of the in vitro studies we have performed previously. Kinetic analyses may be another way to identify patients with different levels of risk from this disease and thereby provide an additional prognostic parameter. This information may also help to individualize future therapies for specific patients based on the in vivo biology in their particular B-CLL clone.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Chiorazzi, MD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute for Medical Research, Manhasset, New York, United States